CLINICAL TRIAL: NCT05928416
Title: ALS Diagnosis From a Saliva Sample: a Non-coding RNA Analysis Approach
Acronym: RNALS
Status: Recruiting | Type: Observational
Sponsor: ZIWIG (Industry)
Collaborators: Monitoring Force Group (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-01
Record Dates: First submitted 2023-06-23; First posted 2023-07-03 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Amyotrophic Lateral Sclerosis, Sporadic; Amyotrophic Lateral Sclerosis
Keywords: ALS; RNA; Saliva sample
MeSH Terms: conditions — Amyotrophic lateral sclerosis 1; Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SLA group: 300 patients
  Interventions: Diagnostic Test: Saliva sample
- Control group: 300 patients
  Interventions: Diagnostic Test: Saliva sample

INTERVENTIONS:
Diagnostic Test: Saliva sample — During the inclusion visit :
  * a neurological examination is taken
  * a saliva sample is taken
  Groups: Control group
Diagnostic Test: Saliva sample — During the inclusion visit :
  * a saliva sample is taken
  Groups: SLA group

SUMMARY:
RNALS is a multicentre, transversal, diagnostic and non-interventional study carried out in ALS reference centers; in order to identify a diagnostic signature for Amyotrophic Lateral Sclerosis by analyzing of coding and non-coding RNA contained in patients saliva.

The study population consists of patients with definite or probable amyotrophic lateral sclerosis (ALS) according to the El Escorial criteria ("ALS Subjects" group) and subjects with no neurological history (Control group).

The control group will be made up of caregivers of patients with ALS, and caregivers of patients with a pathology other than ALS.

The ALS patients concerned by the study already benefit from routine medical care in ALS expert centers in France.

The patients concerned by the study will be managed without modification of the care pathway, nor modification of the therapeutic indications, nor modification of the diagnostic or follow-up examinations necessary according to the context, which are carried out according to the recommendations of the HAS, CNGOF.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age,
* Patient from one of the 2 study populations:

  * Diagnosis of definite or probable ALS according to El Escorial criteria ("patients ALS" group) ;
  * Control group
* Patient able to carry out a mouth rinse,
* Patient affiliated to the healthcare system,
* Patient has dated and signed the consent form,

Exclusion Criteria:

* Recent (<1 month) or ongoing bacterial or viral infection,
* Known active oral or digestive mycosis,
* Evolving, symptomatic or obvious oral pathology,
* Known pregnancy,
* Patient participating in another clinical research study,
* Patient deprived of liberty by administrative or judicial decision or under guardianship ;
* Subject refusing to take a saliva sample;
* For the control group: direct relationship (siblings, descendants, ascendants) with a patient included in the study;
* For control group: medical history of neurological disease (excluding migraine).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be made up with amyotrophic lateral sclerosis (ALS) patients defined or probable according to El Escorial criteria ("ALS patients" group) and patients with no medical history or neurological symptoms (Control Group).
  The control group will be made up of people accompanying the patients (with or without ALS).
  The ALS patients in the study already benefit from routine medical care in ALS expert centers in France. .
  The patients concerned by the study are managed without modification of the care pathway, no modification of the therapeutic indications, no modification of the diagnostic examinations or follow-up necessary according to the context, which are carried out according to the recommendations of the HAS.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-07-11 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC) of the Receiver Operating Curve (ROC) | Through the end of study inclusions, an average of 2 years
  Identify a diagnostic signature for Amyotrophic Lateral Sclerosis by analyzing of coding and non-coding RNA contained in the saliva.

CONTACTS AND LOCATIONS:
Locations (19):
- France (19):
  - CHU Strasbourg, Strasbourg, Alsace
  - CHU Nantes, Saint-Herblain, Loire-Atlantique
  - C.H.U. de Saint-Étienne, Saint-Étienne-de-Montluc, Pays de la Loire Region
  - Hospices Civils de Lyon, Bron, Rhône
  - CHU Angers, Angers
  - CHU Bordeaux, Bordeaux
  - Hôpital Cavale Blanche, Brest
  - CHU Caen, Caen
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHRU Lille, Lille
  - CHU Dupuytren, Limoges
  - Hôpital de La Timone, Marseille
  - CHU Montpellier, Montpellier
  - CHU Nice, Nice
  - Hôpital de la Pitié-Salpêtrière, Paris
  - CHU Rennes, Rennes
  - CHU de la Réunion, Saint-Pierre
  - CHU Toulouse, Toulouse
  - CHU Bretonneau, Tours